CLINICAL TRIAL: NCT04724954
Title: Arm Motor Rehabilitation, Entertainment and Cognition System for the Elderly
Brief Title: Arm Motor Rehabilitation, Entertainment and Cognition System for the Elderly (Clinical Trial)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bright Cloud International Corp (Industry)
Collaborators: Kessler Foundation (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Grigore Burdea, Chief Technology Officer, Bright Cloud International Corp
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Phase IIB Clinical Trial; R44AG044639 (NIH)
Record Dates: First submitted 2021-01-12; First posted 2021-01-26 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Acute Stroke
Keywords: acute stroke; sub-acute stage
MeSH Terms: conditions — Stroke | interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: Number of subjects: The Investigators expect to enroll up to 40 subjects, inpatients and then outpatients at a research hospital and its outpatient clinic at Kessler Foundation: 20 stroke patients, and 20 will be their spouses/caregivers of subjects participating in the randomized control trials component of this study.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Rehabilitation Therapy on Experimental Robotic Table and standard of care (Experimental): 10 elderly 5 days or more post-CVA admitted to Kessler Institute for Rehabilitation/Kessler Foundation) for inpatient rehabilitation will be recruited for experimental group.
  The investigators will also recruit the 10 caregivers of the experimental subjects. Both experimental and control groups will undergo standardized evaluations for motor function/impairment, cognition and emotive states.
  Interventions: Device: Rehabilitation Therapy on Experimental Robotic Table and standard of care
- Rehabilitation Therapy as part of Standard of Care (Sham Comparator): 10 elderly 5 days or more post-CVA admitted to Kessler Institute for Rehabilitation/Kessler Foundation) for inpatient rehabilitation will be recruited as a control group.
  The investigators will also recruit the 10 caregivers of the control subjects. Both experimental and control groups will undergo standardized evaluations for motor function/impairment, cognition and emotive states.
  Interventions: Genetic: Rehabilitation Therapy as part of Standard of Care (Control)

INTERVENTIONS:
Device: Rehabilitation Therapy on Experimental Robotic Table and standard of care — Experimental group will receive VR game-based rehabilitation therapy through Bright Cloud's proprietary device, called BrightArm Compact (BAC). They will also receive Standard of Care rehabilitation
  Other Names: BrightArm Compact Rehabilitation
  Arms: Rehabilitation Therapy on Experimental Robotic Table and standard of care
Genetic: Rehabilitation Therapy as part of Standard of Care (Control) — Control group will receive Standard of Care training only
  Arms: Rehabilitation Therapy as part of Standard of Care

SUMMARY:
The research project is intended to provide information pertaining to the usability, feasibility and clinical benefit of the BAC system for early sub-acute post CVA rehabilitation, improved cognition and emotive state while in acute inpatient rehabilitation settings (Kessler Foundation) and in an outpatient clinic at the same research hospital.

The randomised controlled trials will take place at Kessler Foundation (West Orange, NJ). It will develop a new longitudinal therapy for elderly stroke survivors who are inpatients and then outpatients at a regional rehabilitation hospital, by adding BAC training to customary care for both inpatients and outpatients. Two systems will be used, improving continuity of care (one each for inpatient and outpatient settings).

DETAILED DESCRIPTION:
This study targets participants, who had suffered a stroke very recently, who may or may not have been diagnosed with mild cognitive impairments or dementia (including Alzheimer's disease). It is important to find out if these improvements can be obtained with the computer game-based integrative (motor-cognitive) bimanual rehabilitation developed by Bright Cloud International Corp, and if these gains transfer to daily activities. The study also aims at determining benefit of continuum care training on the BAC in addition to conventional rehabilitation for participants who are inpatients and then outpatients at a rehabilitation hospital and clinic.

Specific aims are:

BAC technology acceptance (all groups); improved motor function for upper extremity; strengthening shoulder and fingers increased range of motion for arms and fingers; improved independence in activities of daily living; improved cognition; improved emotive state; reduction in perceived upper body pain.

Another component of the research project is a small pilot targeting individuals with Parkinson's disease. For them the project is going to:

determine technology acceptance when using the BrightBrainer system; benefit to arms motor function and strengthening when playing BCI therapeutic games; benefit to reduction or tremor when playing games; cognitive benefits improvement in their well-being.

ELIGIBILITY:
Inclusion Criteria (general)

* Age 50 to 85;
* Healthy age-matched volunteers
* diagnosis of CVA that occurred more than 5 days prior and less than 21 days prior (for the stroke survivors group);
* English speakers;
* UE unilateral or bilateral involvement (from new bilateral CVA)
* motor involvement (FMA score 20 to 45);
* ability to actively move UE more than 10o for shoulder and elbow flexion/extension;
* ability to actively extend fingers at least 5o
* cognitive skills to participate (Montreal Cognitive Assessment (MoCA) [Nasreddine et al 2005] score 10-30).
* The adaptive nature of BBC system hardware and therapeutic games can compensate for the motor limitations due to other co-morbidities. Therefore potential participants will not be excluded due to co-morbidities such as Parkinson or arthritis.

Subjects may have normal cognition, MCI or dementia, since the games can compensate for diminished cognition through built-in cues and instructions.

* Inclusion Criterion for the controlled clinical trials arm at Kessler Foundation

  • Living within 25 miles radius of Kessler Foundation West Orange location. This will facilitate participation in the outpatient clinic training, which follows inpatient rehabilitation.
* Exclusion Criteria. (general)

  * being younger than 50 or older than 85 years of age
  * previous stroke
  * Stroke that occurred more than 20 days prior to enrolment
  * Inability to actively extend fingers at least 5 degrees; v. 7/8/2018
  * Fugl-Meyer scores of 19 or less;
  * severe visual neglect or legally blind
  * severe hearing loss or deafness
  * receptive aphasia or severe expressive aphasia;
  * severe spasticity (Modified Ashworth Scale 4/4)
  * contractures of the upper limb joints
  * uncontrolled hypertension (>190/100 mmHg)
  * severe cognitive impairment determined by Montreal Cognitive Assessment (MoCA) [Nasreddine et al, 2005] test of 9 and below;
  * No chemodenervation or nerve block to upper limb involved during the experimental period (e.g., botulinum toxin injection)
  * inability to speak English;
  * a history of violence or drug abuse.
  * paranoia and psychotic behaviour.
  * inability participate in the neuropsychological pre-study assessment for reliable scores (e.g., cognitive impairment, communication disorders).

Exclusion Criteria. (Controlled study arm)

o Those living outside approximately 25 miles radius of Kessler Foundation West Orange location. Those living too far will have a harder time completing the study as outpatients, as they will probably choose clinics closer to home.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Fugl-Meyer Assessment score for upper extremity function (UE sub-set) | Change between baseline, at 3 weeks and at 5 weeks post enrollment
  Upper Extremity Mobility and function. It is scored from 0 (minimum score) to 66 (maximum). The higher the score, the better, with 66 indicating normal upper extremity function.
Change in Cognitive executive function assessment score | Change between baseline, at 3 weeks and at 5 weeks post enrollment
  Trail Making Test B (TMT-B), Neuropsychological Assessment Battery (NAB) Executive Functioning Module. This is a timed test (seconds) with less time indicative of better executive function. No scale.

SECONDARY OUTCOMES:
Change in Arm Range of Motion | Change between baseline, at 3 weeks and at 5 weeks post enrollment
  Measurement of active movement range for shoulder, elbow, and wrist. Measured with a mechanical goniometer, higher angular values indicating larger movement range.
Change in Grasp strength for whole hand (power grasp) and finger pinch | Change between baseline, at 3 weeks and at 5 weeks post enrollment
  Grasp strength and pinch strength measurements using dynamo-meter and pinch meter, respectively. Measured three times for maximal exertion, then averaged. Higher values are better, indicating less hand weakness.
Change in Finger Range of Motion measured with mechanical goniometer | Change between baseline, at 3 weeks and at 5 weeks post enrollment
  finger extension/flexion range for proximal-metacarpal joints. Measured with mechanical goniometer
Change in Upper extremity functional index (UEFI-20) of independence in activities of daily living | Change between baseline, at 3 weeks and at 5 weeks post enrollment
  Self report of degree of independence in activities of daily living (ADLs). Consists of 20 questions, each scored on a 5 point scale with 0 complete dependence (unable to perform task) to 4 independence in a tasks. Minimum score is 0 (subjects is unable to perform any of the 20 listed tasks to 80 complete independence in all 20 ADLs. Higher score is better outcome.
Change in Stroke Impact Scale (SIS) measuring impact of stroke on independence in daily activities | Change between baseline, at 3 weeks and at 5 weeks post enrollment
  Self report of degree of independence in activities of daily living (ADLs). Consists of questions, each scored on a 5 point Likert scale with 1 complete dependence (unable to perform task) to 5 independence in a tasks. Minimum score is 0 (subjects is unable to perform any of the 20 listed tasks to 80 complete independence in all 20 ADLs.
Change in CAHAI 9 Score of independence in bimanual ADLs | Change between baseline, at 3 weeks and at 5 weeks post enrollment
  Chedoke Arm and Hand Activity Inventory, reflecting ADL independence in simulated bimanual ADLs. It consists of 9 tasks, each scored from 1 to 7, where 1 indicates need for total assistance (typical of very weak arms) to 7 indicating total independence in the task. Score range is 9 (minimum) to 63 (maximum)
Game % Score (baseline and performance) in therapeutic games | through study completion, an average 5 weeks from enrollment
  BrightBrainer game performance %, with each game being scored individually. Scores converted to % of task achieved with range of 0% (worst outcome) to 100% (best outcomes).
Game difficulty levels | through study completion, an average 5 weeks from enrollment
  BrightBrainer game difficulty settings, indicating game play intensity and challenge. Each game has levels from 1 (easiest) to 10 (hardest). Higher difficulty the subjects is able to play a game at represents a better outcome.
Average game difficulty levels per session | through study completion, an average 5 weeks from enrollment
  BrightBrainer game difficulty averaged for all games played in a session. Higher average difficulty is indicative of higher function with 1 (easiest) to 10 (hardest). Higher average game difficulty represents a better outcome.
Participants' feedback through subjective evaluation of the system | at 3 weeks and at 5 weeks post enrollment
  Subject feedback and overall ratings on BrightBrainer games, rated on a Likert scale with 1 being least desirable (strongly disagree) to 5 being most desirable rating (strongly agree).
Change in Verbal attention as measured by the Neuropsychological Assessment Battery | Change between baseline, at 3 weeks and at 5 weeks post enrollment
  Attention module digit span tests verbal attention when subject is spoken a sequence of digits, then asked to repeat that sequence. Subjects is spoken 10 sequences of increasing length of digits (between 1 and 9). Score is 1 if sequence is repeated correctly, 0 otherwise. Min score 0 means no spoken digit sequence was repeated correctly, 10 is maximum score, all sequences were repeated correctly by subject.
Change in visual attention as measured by Neuropsychological Assessment Battery | Change between baseline, at 3 weeks and at 5 weeks post enrollment
  Visual attention measured with the dots test of the Neuropsychological Assessment Battery (NAB). This is a delayed recognition span paradigm, in which an array of dots is exposed for a brief period, followed by a blank interference page, followed by a new array with one additional dot. The subject needs to point to the "new" dot. Test administered 3 times, minimum score 0 (none of the new dots found) to maximum 3 (all 3 new dots found).
Change in Beck Depression Inventory II (BDI II) score, a measure of depression severity | Change between baseline, at 3 weeks and at 5 weeks post enrollment
  participants' depression measure with higher scores indicating higher severity (worse mood). Score range is 0 to 63, with 0 indicating normal mood (no depression), 1-13 minimal depression, 14-19 mild depression, 20-28 for moderate and 29-63 severe depression.
Caregiver evaluation of experimental system | at 5 weeks from enrolment
  Rating of system perceived benefit to the person the caregiver cares for. Rating uses a Likert scale with 1 being least desirable outcome and 5 most desirable one.

OTHER OUTCOMES:
Change in Verbal memory as measured by Hopkins Verbal Learning Test, Revised | Change between baseline, at 3 weeks and at 5 weeks post enrollment
  Hopkins Verbal Learning Test, Revised (HVLT-R) is a measure of verbal memory. It provides a brief assessment of immediate recall, delayed recall and delayed recognition. Subject is read a series of nouns in several categories, and the asked t repeat these nouns by writing them on a piece of paper. The test is repeated three times, and each time the score is a count of how many nouns were remembered by the subject. The second phase of the test involves delayed recall, which is administered after about 20 minutes from the original test. subject needs to write down all the nouns they remembered and these are counted. There is a maximum of 12 correct responses during delayed recall, so max score is 12
Change in visuospatial memory as measured by Brief Visuospatial Memory Test, Revised (BVMT-R) | Change between baseline, at 3 weeks and at 5 weeks post enrollment
  Brief Visuospatial Memory Test, Revised (BVMT-R) is a measure of visuospatial memory. In three Learning Trials, the subject views a stimulus page showing an geometric figure for 10 seconds, and there are 6 drawings presented. Then the subject is asked to draw as many of the figures as possible in their correct location on a page in the response booklet. A Delayed Recall Trial is administered after a 25-minute delay. Last, a Recognition Trial, in which the respondent is asked to identify which of 12 figures were included among the original geometric figures, is administered. Raw scores will be used, with higher numbers representing better outcomes. Raw score range is 0 (worst outcome) to 6 (best outcome)
Change in cognitive function as measured by the Montreal Cognitive Assessment Test score | Change between baseline, at 3 weeks and at 5 weeks post enrollment
  Montreal Cognitive Assessment (MoCA) is a standardized test of cognitive function. It consists of question in several cognitive domains and has a maximum score of 30. Cognitive function is considered normal for scores above 26, with scores below 18 being indicative of severe cognitive impairments. Higher score is better.
Change in score for Boston Naming Test of naming objects | Change between baseline, at 3 weeks and at 5 weeks post enrollment
  Boston naming test uses line drawings of objects of graded difficulty. Subject is ask to name (i.e. find nouns associated with) the object depicted in the line drawings. Scoring is based on how many objects (out of 80) were correctly named. Higher score means better cognitive function.
Blood pressure measured with medical meter | through study completion, an average 5 weeks from enrollment
  Systolic and Diastolic Blood pressures measured before, mid way and at end of every experimental session.
Heart rate measured with medical meter | through study completion, an average 5 weeks from enrollment
  Heart rate measured before, mid way and at end of every experimental session.

CONTACTS AND LOCATIONS:
Overall Officials: Grigore C Burdea, PhD, Study Director — Bright Cloud International Corp
Locations (2):
- United States (2):
  - Bright Cloud Int'l Corp, North Brunswick, New Jersey
  - Kessler Foundation, West Orange, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BCI's corporate site showing therapeutic games used with the device — http://www.BrightBrainer.com